CLINICAL TRIAL: NCT00898482
Title: Pancreatic Cancer Serum and Peripheral Blood Lymphocyte Repository
Brief Title: Collecting and Storing Samples of Blood From Patients With Pancreatic Cancer and Healthy Participants
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: JHOC-J0533 CDR0000452792; P30CA006973 (NIH); JHOC-J0533; JHOC-05042601
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy individuals
  Interventions: Other: This is a non-intervention study for all groups.; Other: study of socioeconomic and demographic variables
- At risk individuals
  Interventions: Other: This is a non-intervention study for all groups.; Other: study of socioeconomic and demographic variables
- Cancer patients
  Interventions: Other: This is a non-intervention study for all groups.; Other: study of socioeconomic and demographic variables

INTERVENTIONS:
Other: This is a non-intervention study for all groups. — This is a non-intervention study.
Other: study of socioeconomic and demographic variables — Non-intervention study.

SUMMARY:
RATIONALE: Collecting and storing samples of blood from patients with cancer and healthy participants to test in the laboratory may help the study of cancer in the future.

PURPOSE: This study is collecting and storing samples of blood from patients with pancreatic cancer and healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish a central pancreatic cancer specimen (including serum and peripheral blood lymphocytes) repository to serve as a resource for current or future scientific studies.
* Utilize the clinical database to perform clinicopathologic correlation with the results of those studies.
* Test new hypotheses as they emerge.

OUTLINE: This is a prospective study.

Blood is collected from patients with pancreatic cancer at baseline and then every 3-6 months for up to 2 years. All other participants have blood collected at baseline and complete questionnaires at baseline and then every 3-6 months for up to 2 years. Serum and peripheral blood lymphocytes obtained from the blood samples are frozen and stored.

PROJECTED ACCRUAL: A total of 200 patients and 200 other participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Histologically confirmed pancreatic malignant neoplasm
  * Serologically or image-confirmed diagnosis of pancreatitis or nonmalignant pancreatic disease
  * Healthy, at-risk participant meeting the following criteria:

    * Smoker, diabetic, and/or has a family history of pancreatic cancer
  * Healthy participant (no history of cancer)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The three cohorts are: 1) Healthy individuals, 2) At risk individuals and 3) Cancer patients.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2005-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Establishment of a central pancreatic cancer specimen repository | No time frame
Utilization of the clinical database to perform clinicopathologic correlation with the results of current or future scientific studies | No time frame
Test new hypotheses as they emerge | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Laheru, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins